CLINICAL TRIAL: NCT05129644
Title: Phase I, Randomized Double-Blind, Active Control, Single Dose Escalation Study of P1101 in Healthy Adult Male Subjects
Brief Title: Single Dose Escalation Study of P1101 in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: A09-102
Record Dates: First submitted 2021-11-02; First posted 2021-11-22 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteers
Keywords: P1101, phase 1, healthy volunteers
MeSH Terms: interventions — peginterferon alfa-2a

STUDY DESIGN:
Intervention Model Description: This was a single center, double-blind, randomized, active control, single dose escalation study, with P1101 (24, 48, 90, 180, 225, 270 mcg) as the test drug and Pegasys (180 ug) as the control drug.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- P1101 24 mcg (Experimental): A total of 6 subjects received single dose of 24 mcg P1101
  Interventions: Drug: P1101 (24 mcg)
- P1101 48 mcg (Experimental): A total of 6 subjects received single dose of 48 mcg P1101
  Interventions: Drug: P1101 (48 mcg)
- P1101 90 mcg (Experimental): A total of 6 subjects received single dose of 90 mcg P1101
  Interventions: Drug: P1101 (90 mcg)
- P1101 180 mcg (Experimental): A total of 6 subjects received single dose of 180 mcg P1101
  Interventions: Drug: P1101 (180 mcg)
- P1101 225 mcg (Experimental): A total of 6 subjects received single dose of 225 mcg P1101
  Interventions: Drug: P1101 (225 mcg)
- P1101 270 mcg (Experimental): A total of 6 subjects received single dose of 270 mcg P1101
  Interventions: Drug: P1101 (270 mcg)
- Pegasys 180 mcg (Active Comparator): A total of 12 subjects received single dose of 180 mcg Pegasys
  Interventions: Drug: Pegasys

INTERVENTIONS:
Drug: P1101 (24 mcg) — P1101 solution for injection, 180 mcg/mL, 1.2 mL/vial;Dose/subject: 24 mcg subcutaneously.
  Arms: P1101 24 mcg
Drug: P1101 (48 mcg) — P1101 solution for injection, 180 mcg/mL, 1.2 mL/vial;Dose/subject: 48 mcg subcutaneously.
  Arms: P1101 48 mcg
Drug: P1101 (90 mcg) — P1101 solution for injection, 180 mcg/mL, 1.2 mL/vial;Dose/subject: 90 mcg subcutaneously.
  Arms: P1101 90 mcg
Drug: P1101 (180 mcg) — P1101 solution for injection, 180 mcg/mL, 1.2 mL/vial;Dose/subject: 180 mcg subcutaneously.
  Arms: P1101 180 mcg
Drug: P1101 (225 mcg) — P1101 solution for injection, 180 mcg/mL, 1.2 mL/vial;Dose/subject: 225 mcg subcutaneously.
  Arms: P1101 225 mcg
Drug: P1101 (270 mcg) — P1101 solution for injection, 180 mcg/mL, 1.2 mL/vial;Dose/subject: 270 mcg subcutaneously.
  Arms: P1101 270 mcg
Drug: Pegasys — Pegasys for injection, 180 mcg/mL, 1.0 mL/vial, Dose/subject: 180 mcg subcutaneously.
  Other Names: peginterferon alfa-2a
  Arms: Pegasys 180 mcg

SUMMARY:
This was a single-center, double-blind, randomized, active control, single dose escalation study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) profiles of P1101 in 48 healthy volunteers.

DETAILED DESCRIPTION:
The primary objectives were to determine the safety and tolerability of single ascending subcutaneous doses of P1101 and to determine the pharmacokinetics of P1101 in single ascending subcutaneous doses of P1101 in healthy male subjects.

The secondary objectives were to evaluate the occurrence of side effects in healthy subjects receiving either P1101 or PEGASYS; to compare the pharmacokinetic parameters for P1101 and PEGASYS; and to assess the effect of P1101 on the biomarkers 2',5' oligoadenylate synthetase and neopterin.

A total of 48 subjects were enrolled to receive subcutaneous injection of P1101 in the dose level of 24 , 48 , 90 , 180 , 225 , or 270 mcg or to receive subcutaneous injection of 180 mcg Pegasys.

ELIGIBILITY:
Main Inclusion Criteria:

1. Be healthy males, non-smokers, ≥18 and ≤45 years of age;
2. Able to attend all scheduled visits and to comply with all study procedures.

Main Exclusion Criteria:

1. Clinically significant illness or surgery within 4 weeks prior to dosing;
2. Any clinically significant abnormality or abnormal laboratory test results found during screening;
3. Positive test for hepatitis B, hepatitis C, or HIV at screening;
4. Clinically significant vital sign abnormalities at screening;
5. History of significant alcohol or drug abuse within one year prior to the screening visit;
6. History of severe allergic or hypersensitivity reactions;
7. Use of an investigational drug or participation in an investigational drug trial within the last 4 weeks;
8. Any clinically significant history or presence of neurological, cardiovascular, pulmonary, hematological, immunologic, metabolic or other uncontrolled systemic disease;
9. Clinically significant history or known presence of psychiatric disorders, including but not limited to depression, anxiety, and sleep disorders;
10. Body organ transplant and are taking immunosuppressants;
11. History of malignant disease;
12. History or presence of endocrine disorders;
13. History of coagulation disorders and blood dyscrasias;
14. Inability to comprehend the written consent form.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-11-07 (Actual); Primary Completion 2010-06-26 (Actual); Study Completion 2010-06-26 (Actual)

PRIMARY OUTCOMES:
Adverse Event | Through study Day 35
  Frequency and severity of all adverse events among subjects, including frequency and severity of drug-related adverse events.
AUC of P1101 and Pegasys | Samples were collected within 1 hour pre-dose, and at 1, 3, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192, 240, 288, 336, 504, and 672 hours post-dose.
  Area under the serum concentration-time curve from time 0 to infinity
AUC0-t of P1101 and Pegasys | Samples were collected within 1 hour pre-dose, and at 1, 3, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192, 240, 288, 336, 504, and 672 hours post-dose.
  Area under the serum concentration-time curve from time zero to the last measurable concentration (AUC0-t)
Cmax of P1101 and Pegasys | Samples were collected within 1 hour pre-dose, and at 1, 3, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192, 240, 288, 336, 504, and 672 hours post-dose.
  Maximum serum concentration; the highest concentration observed during a dosage interval.
Ct of P1101 and Pegasys | Samples were collected within 1 hour pre-dose, and at 1, 3, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192, 240, 288, 336, 504, and 672 hours post-dose.
  The last measured serum concentration, the last concentration above the lower limit of quantification following dose
Tmax of P1101 and Pegasys | Samples were collected within 1 hour pre-dose, and at 1, 3, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192, 240, 288, 336, 504, and 672 hours post-dose.
  The time that Cmax was observed
T½ of P1101 and Pegasys | Samples were collected within 1 hour pre-dose, and at 1, 3, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192, 240, 288, 336, 504, and 672 hours post-dose.
  Terminal elimination half-life
λz (Ke) of P1101 and Pegasys | Samples were collected within 1 hour pre-dose, and at 1, 3, 6, 9, 12, 16, 24, 36, 48, 72, 96, 120, 144, 168, 192, 240, 288, 336, 504, and 672 hours post-dose.
  The terminal elimination rate constant; calculated using linear regression on the terminal portion of the Ln-concentration versus time curve

SECONDARY OUTCOMES:
2',5' oligoadenylate synthetase (OAS): Emax | Samples were collected within 1 hour pre-dose and at 24, 48, 72, 96, 120, 168, 240, 336, 504, and 672 hours post-dose
  Maximum serum biomarker response; the highest biomarker concentration observed during a dosage interval.
2',5' oligoadenylate synthetase (OAS): Tmax | Samples were collected within 1 hour pre-dose and at 24, 48, 72, 96, 120, 168, 240, 336, 504, and 672 hours post-dose
  The time that Emax was observed.
2',5' oligoadenylate synthetase (OAS): AUC0-t | Samples were collected within 1 hour pre-dose and at 24, 48, 72, 96, 120, 168, 240, 336, 504, and 672 hours post-dose
  Area under the biomarker concentration versus time curve from time 0 to the last measured concentration.
Neopterin: Emax | Samples were collected within 1 hour pre-dose and at 24, 48, 72, 96, 120, 168, 240, 336, 504, and 672 hours post-dose
  Maximum serum biomarker response; the highest biomarker concentration observed during a dosage interval.
Neopterin: Tmax | Samples were collected within 1 hour pre-dose and at 24, 48, 72, 96, 120, 168, 240, 336, 504, and 672 hours post-dose
  The time that Emax was observed.
Neopterin: AUC0-t | Samples were collected within 1 hour pre-dose and at 24, 48, 72, 96, 120, 168, 240, 336, 504, and 672 hours post-dose
  Area under the biomarker concentration versus time curve from time 0 to the last measured concentration.

OTHER OUTCOMES:
Immunogenicity | Samples were collected within 1 hour pre-dose, at 336 and 672 hours after dose administration
  Analysis of the concentration of anti-P1101 antibody.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, MD, Principal Investigator — Anapharm 5160, boul. Décarie, suite 800 Montréal, Québec, Canada, H3X 2H9
Locations (1):
- Anapharm, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang YW, Qin A, Fang J, Wang TF, Tsai CW, Lin KC, Teng CL, Larouche R. Novel long-acting ropeginterferon alfa-2b: Pharmacokinetics, pharmacodynamics and safety in a phase I clinical trial. Br J Clin Pharmacol. 2022 May;88(5):2396-2407. doi: 10.1111/bcp.15176. Epub 2021 Dec 28. PMID 34907578